CLINICAL TRIAL: NCT04298632
Title: Reducing Pesticide Exposure Among Latino Adolescents Through a Promotora-based Intervention
Brief Title: Latino Youth Agricultural Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska Lincoln (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 20734; 2U54OH007541-16 (NIH)
Record Dates: First submitted 2020-03-03; First posted 2020-03-06 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Pesticide Safety
Keywords: Latino Youth

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Youth-only (Experimental): Only the youth receives the education program
  Interventions: Behavioral: Safety Education Program
- Family enhanced (Experimental): A parent and the youth both receive the education program
  Interventions: Behavioral: Safety Education Program
- Control (No Intervention): neither parent, nor youth receives the education program

INTERVENTIONS:
Behavioral: Safety Education Program — this is a pesticide safety education program
  Arms: Family enhanced; Youth-only

SUMMARY:
This project implements and evaluates a promotora-based intervention targeted at adolescent farm workers. The goal of the project is to determine the effectiveness of each intervention in promoting increased knowledge and practice of pesticide safety behaviors.

DETAILED DESCRIPTION:
This project implements and evaluates a promotora-based intervention targeted at adolescent farm workers. The intervention will be delivered to two different treatment groups: 1) adolescent only, adolescents receive the adapted adolescent version of La Familia Sana program and 2) family enhanced, adolescent and mother both receive the La Familia Sana program. In addition, there will be a control group where adolescent farmworkers will not be exposed to any pesticide safety program. Our project will:

1. Determine if a promotora-based intervention targeting pesticide safety in the workplace is effective in increasing knowledge about safety behaviors among Latino adolescents engaged in farm work.
2. Delineate variation by group among adolescents' knowledge about safety behaviors.
3. Delineate variation in adolescents' pesticide safety behaviors and neurological outcomes after intervention between all groups.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent self-identifies as Latino, Hispanic, or of Latin American heritage
* Adolescent is between the ages of 12-21
* Adolescent has been engaged (paid or unpaid) in farm work for at least 10 hours in he last 30 days
* Adolescent has a parent living with them

Exclusion Criteria:

* Refusal of youth to provide assent or parent to provide consent

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 118 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
knowledge of pesticide safety behaviors | 7 weeks
  This outcome measure will be assessed by a series of nine questions asking adolescents "How do you believe that farmworkers can come in contact with pesticides while working?" Additionally, nine additional questions will be asked that assess "How do you believe that farmworkers can have contact with pesticides while at home?" All responses for these questions are "yes" or "no"
Self-protective behaviors | 7 weeks
  Self-protective behaviors will be assessed by items asking adolescents about their clothes wearing and handling and their hand washing behaviors. Items regarding clothes wearing and handling include self-reported frequency of removing shoes and clothes prior to entering their home and wearing the same clothes more than one day. Additionally, several questions ask about the frequency of wearing shorts, sandals, gloves, etc. Regarding hand washing behavior, adolescents will self-report their hand washing behaviors at pretest and posttest. These questions ask youth about the frequency in which they wash their hands prior to eating, drinking, chewing gum, using the restroom, touching co-workers, etc. All self-protective behavior questions have a response option of "never", "sometimes", "usually", and "always"

SECONDARY OUTCOMES:
Neurological functioning | 7 weeks
  Neurological functioning in the form of coordination and fine motor skills will be assessed by the finger tapper test. This measure focuses specifically on speed and is sensitive to the effects of neurotoxicants. The finger tapper test produces a mean score for both the participant's dominant and non-dominant hand as a result of a series of 10 second tapping exercises.

CONTACTS AND LOCATIONS:
Locations (1):
- Oklahoma State University, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes
The data collected from this project will be made available to other researchers within 2 years of completing the project. Those wishing to use the data will be required to submit an application indicating the purpose for which the data will be used and documenting that the research protocol has been approved by the appropriate IRB. Any costs involved in the providing access to data (e.g., statistical and programming support, duplication of documentation) will be paid by those requesting access.
Supporting Information: Study Protocol, ICF
Time Frame: Data will become available within 2 years of completing the project and be available for up to five years.
Access Criteria: Those wishing to use the data will be required to submit an application indicating the purpose for which the data will be used and documenting that the research protocol has been approved by the appropriate IRB.